CLINICAL TRIAL: NCT05412901
Title: Scaffolding of Brain Operations: the Role of Beta Oscillations in Forming Flexible Neural Ensembles
Brief Title: Scaffolding of Brain Operations
Acronym: BETATEST
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: In response to quality assurance and compliance concerns about some specific studies, NYSPI is undertaking an Institute-wide safety review of human subjects research protocols. HHS OHRP issued an FWA restriction on NYSPI research as of 2023/6/23.
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Saskia Haegens, Assistant Professor of Clinical Neuroscience, New York State Psychiatric Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: R01MH123679 (NIH)
Record Dates: First submitted 2022-06-01; First posted 2022-06-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Behavioral Performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Visual spatial discrimination task (Other): exp 1.1
  Interventions: Other: discrimination task
- Visual spatial discrimination task with temporal manipulation (Other): exp 1.2
  Interventions: Other: discrimination task
- Crossmodal discrimination task (Other): exp 3.1
  Interventions: Other: discrimination task
- Visual rule-switching discrimination task [gratings] (Other): exp 3.2
  Interventions: Other: discrimination task
- Visual rule-switching discrimination task [images] (Other): exp 3.3
  Interventions: Other: discrimination task

INTERVENTIONS:
Other: discrimination task — Participants perform a discrimination task while their brain activity is recorded with EEG. Beta power will be estimated using spectral decomposition techniques, zooming in on subject specific bands in temporospatial windows of interest, and correlated with (1) WM content, (2) decision outcome, and (3) behavioral performance (i.e., accuracy and RT).

SUMMARY:
Brain activity will be recorded while participants rest and/or perform perceptual discrimination tasks. These tasks include the presentation of sensory stimuli and require participants to detect and discriminate these stimuli, and to report about the objective properties of the stimuli as well as about their subjective perceptual experience using ratings of confidence, visibility, and/or alertness/sleepiness. All sensory stimuli used are neutral and consist of visual stimuli presented on a computer screen (either basic visual stimuli, e.g. an arrow, a grating or a dot, or neutral pictures of e.g. objects, buildings, landscapes), or auditory stimuli presented via headphones (either basic sounds, e.g. a beep or noise, or more complex sounds, e.g. a spoken word or rhythm). The experimental tasks may require participants to compare between sensory stimuli presented at different spatial locations or at different times, and/or to focus their attention on specific stimuli while suppressing distracting information; additionally, tasks may require participants to remember these stimuli for a delayed report. In these tasks, participants' performance will be quantified by motor responses (i.e., button press), reaction times and subjective ratings (confidence, visibility, alertness/sleepiness).

Brain activity will be recorded by means of electroencephalography (EEG), a non-invasive technique consisting of electrodes placed along the scalp that record electrical field potentials generated by cortical neurons. EEG will be used to record brain activity prior to and in response to the sensory stimuli presented during the cognitive and perceptual tasks as well as during the participants' responses. Additionally, EEG may be used to record brain activity during a baseline resting state, while participants are not engaged in any particular tasks. In particular, the analysis of the EEG signal will focus on event-related brain activity (i.e., in response to the stimuli) such as event-related potentials (ERP), as well as ongoing and spontaneous and/or induced brain activity quantified as oscillations: wave-like signal fluctuations reflecting rhythmic variations of membrane potentials of cortical neurons. In addition, the investigators will use MRI to take an anatomical image of the brain to facilitate localizing the sources of the activity measured with EEG.

DETAILED DESCRIPTION:
The brain constantly makes decisions based on perceptual input as well as internal signals, quickly weighing and processing information, leading to goal-directed behavior. One key aspect crucial to all these processes is communication the transfer of information from one brain network to the next. However, we are only beginning to understand how the brain accomplishes this. Here, the investigators propose to study exactly this question. The overarching goal of this project is to elucidate how the brain sets up the functional neural architecture involved in working memory and decision-making. The investigators argue that brain oscillations in the beta frequency band 1530 Hz play a critical role in forming flexible neural ensembles. The investigators propose a novel theoretical framework, delineating how the beta rhythm flexibly sets up transient networks, linking neuronal circuits that are relevant to current task demands, especially in terms of endogenous information processing e.g., working memory, decision-making. In this view, beta provides the scaffolding for information transfer,routing information through the brain by temporarily connecting relevant nodes such that exchange of information can take place. The investigators propose that the beta rhythm briefly activates a neural ensemble, allowing it to broadcast its message encoded in population spike activity such that it can be efficiently and effectively received. To test this framework, the aim here is to (1) examine the role of beta oscillations in dynamic neural ensemble formation and its relation to behavioral performance, (2) identify the underlying circuit-level physiology of beta-mediated ensemble formation, and (3) establish the generality of beta-mediated ensemble formation and identify non-invasive biomarkers. The investigators will use a combination of EEG recordings in healthy human subjects, and intracranial electrophysiology and optogenetic neuromodulation in awake-behaving rodents. Both human subjects and animals will perform a spatial working-memory paradigm, critically allowing vertical integration across recording levels. Human subjects will additionally perform working-memory tasks in different sensory modalities and at higher levels of abstraction to guarantee generalizability of results, and to allow for identification of biomarkers to be used in future patient studies. This approach is designed to answer core mechanistic questions how are local ensembles formed and how are these modulated Critically, the investigators will determine the effect of these mechanisms on behavior. The project will provide fundamental insights that will set the stage for further detailed investigations in healthy human subjects and patients with impaired beta functioning and cognitive impairment, such as in Parkinson's disease and schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Normal (or corrected-to-normal) vision, normal hearing

Exclusion Criteria:

* Epilepsy, past brain surgery, neurological or psychiatric disorders for which they are on medication

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-04-10 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
EEG spectral beta power | during procedure
  Brain activity will be recorded using 96-channel EEG (BrainVision actiCHamp system, Brain Products). Spectral analysis will be performed using the Matlab-based FieldTrip toolbox, a standard in the field. For all spectral analyses, subject-specific peak frequencies will be estimated to tailor the approach. Beta power will be assessed in a band centered at the individual peak frequency.

SECONDARY OUTCOMES:
behavioral performance: accuracy | during procedure
  Accuracy will be assessed as percentage correct responses on the discrimination task.
behavioral performance: reaction time | during procedure
  Reaction times will be assessed per trial on the discrimination task as response time measured from probe onset.

CONTACTS AND LOCATIONS:
Overall Officials: Saskia Haegens, PhD, Principal Investigator — NYSPI
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided